CLINICAL TRIAL: NCT00899535
Title: The Cancer Genome Atlas (TCGA) Utilizing Z0030 NSCLC Patient Samples
Brief Title: Cancer Genome Study Using Samples From Patients With Stage I or Stage II Non-Small Cell Lung Cancer Treated on Clinical Trial ACOSOG-Z0030
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACOSOG-Z4082; ACOSOG-Z4082; CDR0000617514 (Registry Identifier: NCI Physician Reference Desk)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Lung Cancer
Keywords: adenocarcinoma of the lung; large cell lung cancer; squamous cell lung cancer; stage I non-small cell lung cancer; stage II non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung | interventions — Microarray Analysis; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor samples from patients enrolled on Z0030.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: This research study is looking at the cancer genome using tumor samples from patients with stage I or stage II non-small cell lung cancer treated on clinical trial ACOSOG-Z0030. Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.
  Interventions: Genetic: DNA analysis; Genetic: RNA analysis; Genetic: microarray analysis; Genetic: mutation analysis; Genetic: polymorphism analysis

INTERVENTIONS:
Genetic: DNA analysis
Genetic: RNA analysis
Genetic: microarray analysis
Genetic: mutation analysis
Genetic: polymorphism analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at the cancer genome using tumor samples from patients with stage I or stage II non-small cell lung cancer treated on clinical trial ACOSOG-Z0030.

DETAILED DESCRIPTION:
OBJECTIVES:

* To investigate the clinical relevance of conducting comprehensive molecular analyses on clinically annotated high-quality tumor biospecimens from patients with stage I or II, N0 or N1 (less than hilar) non-small cell lung cancer.

OUTLINE: This is a multicenter study.

Biological specimens are collected from participating clinical sites and analyzed by transcription profiling of RNA and microRNA; detection of DNA copy number changes and chromosomal rearrangements; epigenetic modifications analyses; and sequencing of genomic segments, genes, and regulatory regions to assess sequence variation. Clinical information associated with each specimen donor is also collected.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of non-small cell carcinoma

  * Primary, untreated disease
  * Stage I or II (T1 or T2, N0 or non-hilar N1, M0) disease
  * Any of the following histologies allowed:

    * Squamous cell carcinoma
    * Adenocarcinoma (< 10%)
    * Large cell carcinoma (high-grade)
* Available tumor tissue samples collected on clinical trial ACOSOG-Z0030 and meeting the following criteria:

  * Snap-frozen and stored at a temperature of -80°C or lower
  * Specimens may come from any site within the lung or one that is involved by direct regional extension of tumor from the originating site in the lung
* No regional lymph node or distant metastases
* No recurrent or persistent disease after prior neoadjuvant or adjuvant treatment for lung cancer
* Must have matching frozen samples of normal tissue and blood

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with non-small cell carcinoma previously registered on ACOSOG-Z0030.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2008-10; Primary Completion 2010-10 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Clinical relevance of conducting comprehensive molecular analyses on clinically annotated high-quality tumor biospecimens | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Allen, MD, Study Chair — Mayo Clinic